CLINICAL TRIAL: NCT02274441
Title: Gynaecological Emergencies: Validation of Indicators of Activity and Quality of Care for Creation of a Network Sentinel
Brief Title: Activity and Quality of Care Indicators' for a Sentinel Network Creation
Acronym: URGO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI12027
Record Dates: First submitted 2014-10-08; First posted 2014-10-24 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Obstetrics; Maternal Morbidity; Gynecology; Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is no large-scale data in France or internationally, on the quality of care in gynecological emergencies, or the consequences of delay or misdiagnosis of women's health or on determinants of these delays or misdiagnosis. The creation of a sentinel network for gynecological emergencies could help quantify these links and test strategies to avoid the worst effects by implementing simple diagnostic tools from clinical research.

The network will be designed to promote research in women's health and the emergency reception by focusing on:

(i) Assessment of the quality and organization of care and professional practice for the management of gynecological emergencies.

(ii) The study of severe morbidity and its determinants (iii) comparison of organizational practices and health outcomes of women over time within the same department or between services having substantially the same recruitment (iv) Comparison of organization systems gynecological emergencies departement between different high resource francophone countries (France, Switzerland, Belgium).

(v) The assessment of new diagnostic strategies (sorting or diagnostic aid) or therapeutic derived from clinical research.

DETAILED DESCRIPTION:
Objectives :

* To measure the incidence of the potentially life-threatening gynaecological emergencies (G-PLE) and of the Cases of severe morbidity (SM)
* To analyze the determinants of the SM,
* To validate an objective score of quality

Criterias of evaluation:

* Incidence of the G-PLE and SM cases during one month.
* Reliability and validity of measurements of the indicators of quality of care.

Methodology:

Stage 1: Data acquisition (prospective) within 22 gynaecological emergencies departments.

Stage 2: Sampling and checking of files of patients included at stage 1

Calendar of the research project:

18 months:

* 6 months for the phase of preparation,
* 1 month for the investigation of incidence,
* 5 months for the phase of checking data,
* 6 months of statistical analysis

Statistical Analyzes:

Descriptive statistics of the data. Estimation of the incidence rate of the potentially life-threatening gynaecological emergencies (G-PLE) and of the cases of Severe morbidity (SM) among women consulting for acute pelvic pain.

To construct reliable quality indicators, principal components analysis and Cronbach's α statistics will be performed to determine the underlying dimensions. Construct validity of indicators will be assessed by testing predefined hypotheses about relationship between G-PLE and or SM and quality indicators.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking gynaecological emergencies departments leaned with a public maternity volunteers to take part in the study.
* Sample of files resulting from the principal centers recruiters

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Number of centers :
  22 French-speaking gynaecological emergencies departments leaned with a public maternity
  Number of subjects expected:
  2000 consultations for acute pelvic pain, 200 patients hospitalized for data-gathering stage; 408 records for checking data stage
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of the potentially life-threatening gynaecological emergencies (G-PLE ) | 1 year
Incidence of severe morbidity (SM) cases | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Poissy Saint Germain Hospital, Poissy, France